CLINICAL TRIAL: NCT05326932
Title: An Investigator Initiated and Conducted, Prospective, Multicenter, Randomized Outcome-blinded Study of Treating Mechanical Thrombectomy Exceeding 24 Hours in Patients with Acute Ischemic Stroke Due to Large Vessel Occlusion
Brief Title: Large Artery Occlusion Treated in Extended Time with Mechanical Thrombectomy Trial
Acronym: LATE-MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LATE-MT
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Large vessel occlusion; Mechanical thrombectomy; Extended time; Randomised clinical trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Mechanical thrombectomy to be initiated as soon as possible after randomisation.
  Interventions: Procedure: Mechanical thrombectomy
- Control group (No Intervention): Patients assigned to the control group will avoid treating MT and only receive the standard medical treatment according to local guidelines.

INTERVENTIONS:
Procedure: Mechanical thrombectomy — Subjects in intervention group will receive MT as soon as possible. Investigators and clinicians should strive to reduce delays of pre-surgery procedure and follow the local standard guideline of MT during the operation and perioperative period. All CFDA approved devices are allowed in this trial. Angioplasty and stent placement can be performed at the discretion of the physicians. Base on site experience, the randomization-operation start period should be within 60 minutes.
  Arms: Intervention group

SUMMARY:
A multi-center, prospective, randomized, open-label, adaptive group sequential designed, blinded endpoint assessment (PROBE) clinical trial of endovascular treatment among selected AIS

DETAILED DESCRIPTION:
The LATE-MT trial aims to determine that compared with standard medical care without MT, performing MT in a time window that exceeds 24 hours after last seen well, is superior on the functional outcome in AIS patients due to LVO who have been carefully selected by clinical and imaging criteria. The secondary aims include comparing with standard medical care without MT, to determine whether performing MT exceeding 24 hours of last known well is safe on the risks of any ICH, sICH, and any SAE. Other secondary aims include early improvement in neurological recovery as measured by NIHSS scores at 7 days; successful recanalization rate; imaging measurements of infarct size at 24-48 hours; death or major disability (mRS 3-6); separately on death and disability (mRS 3-5); HRQoL using Euro-QoL EQ-5D questionnaire; utility-weighted modified Rankin scale scores; duration of hospitalization; residence; and hospital service costs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Present 24-72 hours of stroke onset or last seen well
3. Clinical diagnosis of AIS due to anterior circulation LVO (from internal carotid artery (ICA) extracranial segment to middle cerebral artery (MCA) M1 and M2 segment) on brain imaging
4. National Institute of Health stroke scale (NIHSS) ≥6 at randomisation
5. Viable cerebral tissue on computerized tomography perfusion (CTP) or magnetic resonance imaging perfusion (MRP) assessed: infarct core volume <50mL, mismatch ratio ≥1.8 and mismatch volume ≥15mL
6. Written informed consent (by patient or proxy, according to local requirements)

Exclusion Criteria:

Clinical Exclusion Criteria

1. Considered unlikely to benefit from trial (e.g. advanced dementia, major pre-stroke disability (prior modified Rankins scale (mRS) ≥2), high likelihood of early death), as judged by the responsible treating clinician
2. Major co-morbid disease that could interfere with outcome assessments and follow-up (e.g. cancer, severe heart failure, kidney failure)
3. Pregnancy
4. Unable to undergo a CTP or MRP
5. Known allergy to iodine, heparin, anaesthesia, or other definite contraindication to receiving endovascular treatment (EVT) procedure
6. Seizures at stroke onset or before randomization and baseline NIHSS scores cannot be accurately determined
7. Baseline blood glucose of <50mg/dL (2.78 mmol/L) or >400mg/dL (22.20 mmol/L)
8. Baseline platelet count <50,000/uL
9. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with International normalized ratio (INR) >3
10. Severe, sustained hypertension (systolic blood pressure (BP) >220 mmHg or diastolic BP >120 mmHg)
11. Presumed septic embolus, suspicion of bacterial endocarditis
12. EVT attempted after stroke onset
13. Unlikely to participate in follow-up assessments
14. Currently participating in another trial that may affect outcomes.
15. Any other condition that, in the opinion of the investigator will pose a significant hazard to the subject if participating in the trial.

Neuroimaging Exclusion Criteria

1. Intracranial hemorrhage (ICH), including parenchymal hemorrhage, ventricular hemorrhage, subarachnoid hemorrhage, and subdural/exsanguination
2. Evidence of intracranial tumor (except small meningioma)
3. Significant mass effect with midline shift
4. Aortic dissection
5. Intracranial stent implanted in the same vascular territory
6. Any other condition that may affect EVT procedure, like the tortuous vascular path the device is difficult to reach the target position or difficult to recover
7. Occlusions in multiple vascular territories confirmed on Computerized tomography angiography (CTA)/ Magnetic resonance imaging angiography (MRA) (e.g. bilateral MCA occlusions, or an MCA and a basilar artery occlusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional recovery (level of disability) | 90 days
  Shift (improvement) in scores on the modified Rankin scale (mRS). The value range 0-6: higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Neurological impairment | 24 hours and 7 days
  Measured by scores on the National Institute of Health Stroke Scale (NIHSS). The value range 0-42: higher scores mean a worse outcome.
Death or major disability | 90 days
  modified Rankin scale (mRS) 3-6
Separately on death and disability | 90 days
  modified Rankin scale (mRS) 3-5
Health-related Quality of Life (HRQoL) | 90 days
  using EQ-5D. European Quality of Life 5-dimensional questionnaire. The EQ-5D comprises five dimensions of health: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, and anxiety and depression. . EQ-5D-5L, includes five levels of severity for each dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems). The value range 0-100: Higher scores mean a worse outcome.
Utility-weighted modified Rankin scale scores | 90 days
  Utility-weighted modified Rankin scale scores. The value range from 0 to 10: higher scores mean a better outcome.
  Higher scores mean a worse outcome.
Duration of hospitalization | 90 days
  Days of hospitalization
Residence | 90 days
  Days of residence
Hospital service costs | 90 days
  Health economic measurement
Infarct volume on DWI, or CT | 24 hours
  Infarct volume on DWI, or CT if DWI not feasible
Recanalization | 24 hours after MT
  Recanalization confirmed on imaging

OTHER OUTCOMES:
Intracerebral hemorrhage (ICH) | 24 hours and 90 days
  a) symptomatic ICH, based on previous criteria; b) ICH of any type in brain imaging
Death | 7 days and 90 days
  Death
Serious adverse events (SAE) | 90 days
  All SAE during follow-up in all randomized patients

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, PhD, Principal Investigator — The George Institute for Global Health, China; Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to the research office of The George Institute for Global Health, Sydney Australia.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: http://georgeinstitute.org.au